CLINICAL TRIAL: NCT02273726
Title: A Phase 3, Open-Label, Randomized, Active-Controlled Study of the Efficacy and Safety of Roxadustat (FG-4592) in the Maintenance Treatment of Anemia in Subjects With End Stage Renal Disease (ESRD) on Stable Dialysis
Brief Title: Study to Evaluate the Efficacy and Safety of Roxadustat in the Treatment of Anemia in Participants With ESRD on Stable Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Collaborators: Astellas Pharma Europe B.V. (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-4592-064
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Results first posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-09

CONDITIONS: CKD Anemia in Stable Dialysis Patients
Keywords: Anemia; Chronic Kidney Disease; Dialysis; hemodialysis; peritoneal dialysis; hemoglobin; End stage renal disease; Stable Dialysis; erythropoietins; erythropoiesis stimulating agent
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Epoetin Alfa; roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Roxadustat (Experimental): Participants will receive roxadustat tablets, administered orally 3 times weekly (TIW). Initial roxadustat dose will be based on the participant's average prescribed erythropoietin stimulating agent (ESA) dose in the 4 weeks (if on epoetin or darbepoetin or 8 weeks (if on Mircera®) prior to randomization. Dose adjustments will be permitted to maintain a hemoglobin (Hb) level of approximately 11 grams (g)/deciliter (dL). The maximum roxadustat dose is 3.0 milligrams (mg)/kilogram (kg) per dose or 400 mg per administration (whichever is lower).
  Interventions: Drug: Roxadustat
- Epoetin Alfa (Active Comparator): Participants on hemodialysis (HD) will receive epoetin alfa, administered intravenously (IV) TIW and participants on home HD or peritoneal dialysis (PD) will receive epoetin alfa, administered subcutaneously (SC). Initial epoetin alfa dose will be based on the participant's average weekly prescribed ESA dose in 4 weeks prior to randomization if on epoetin or darbepoetin, and average monthly (4-week) prescribed ESA dose in 8 weeks prior to randomization if on Mircera®. In case of a change in route of administration from SC to IV (TIW), the initial dose of IV epoetin alfa will be determined by the investigator per local standard of care (SOC). Dose adjustments will follow the recommendations as per the approved country-specific product label (United States Package Insert [USPI] or Summary of Product Characteristics [SmPC]) or local SOC.
  Interventions: Drug: Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin Alfa — Epoetin alfa will be administered per dose and schedule specified in the arm.
  Arms: Epoetin Alfa
Drug: Roxadustat — Roxadustat will be administered per dose and schedule specified in the arm.
  Other Names: FG-4592
  Arms: Roxadustat

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of roxadustat compared with active control (epoetin alfa) for the maintenance treatment of anemia in participants with ESRD on dialysis.

DETAILED DESCRIPTION:
This study will consist of three study periods as follows:

1. Screening Period of up to 6 weeks (8 weeks if on Mircera)
2. Treatment Period: a minimum of 52 weeks, a maximum of up to 3 years from the date last participant is randomized. Minimum study duration for participants enrolled under Protocol Amendment 1 or 2 may be less than 52 weeks
3. A Follow-up period of 4 weeks.

Participants will be randomized in a 1:1 ratio to receive either roxadustat or epoetin alfa (active control) in an open-label manner.

ELIGIBILITY:
Inclusion Criteria:

* Receiving dialysis for ESRD for ≥3 months. Incident dialysis participants (under Amendment 1 and 2) receiving dialysis for ESRD for ≥ 2 weeks but ≤ 4 months at the time of randomization
* Participants must be on ESA for ≥ 8 weeks prior to screening; incident dialysis participants must be on ESA for ≥ 4 weeks prior to screening.
* Mean of the 3 most recent central lab Hb values during the Screening Period must be ≥ 9.0 g/dL and ≤ 12.0 g/dL (for incident dialysis participants, mean of the 2 most recent Hb values must be ≥ 8.5 g/dL and ≤ 12.0 g/dL); with an absolute difference of ≤ 1.3 g/dL between the highest and the lowest value. Samples are obtained at least 4 days apart (2 days under Amendment 2) and the last Hb value must be within 10 days prior to the randomization visit
* Participants with ferritin level ≥ 100 nanograms (ng)/milliliter (mL) (<100 ng/mL under Amendment 2) or transferrin saturation (TSAT) ≥ 20% (<20% under Amendment 2) at screening may qualify upon receiving iron supplement (per local standard of care)
* Participants with a serum folate and Vitamin B12 ≥ lower limit of normal (LLN) (< LLN under Amendment 2) at screening may qualify upon receiving supplement (per local standard of care)
* Participant's alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are ≤3x the upper limit of normal (ULN), and total bilirubin (TBL) is ≤1.5x ULN at screening
* Participant's body weight is 45 kilograms (kg) to 160 kg.

Exclusion Criteria:

* Participant has received an red blood cell (RBC) transfusion within 8 weeks (4 weeks under Amendment 2) prior to randomization
* Participant has known history of myelodysplastic syndrome or multiple myeloma
* Participant has known inherited disease such as thalassemia or sickle cell anemia or other known causes for anemia other than chronic kidney disease.
* Participant has known hemosiderosis, hemochromatosis, coagulation disorder,or hypercoagulable condition
* Participant has known chronic inflammatory disease that could cause anemia
* Participant has anticipated surgery that is expected to cause blood loss
* Participant has known gastrointestinal bleeding
* Participant has history of chronic liver disease (for example, chronic infectious hepatitis,chronic auto-immune liver disease,cirrhosis, or fibrosis of the liver)
* Participant with New York Heart Association (NYHA) Class III or IV congestive heart failure
* Participant has had a heart attack, stroke, seizure, or a thrombotic/thromboembolic event (for example, deep vein thrombosis or pulmonary embolism) within 12 weeks prior to participating in the study
* Participant has uncontrolled high blood pressure within 2 weeks prior to participating in the study
* Participant has a history of malignancy, except for the following: cancers determined to be cured or in remission for ≥2 years, curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ, or resected colonic polyps.)
* Participant is positive for human immunodeficiency virus (HIV), Hepatitis B surface antigen, or anti-hepatitis C virus antibody
* Participant with prior organ transplant who experience rejection within 6 months or on high doses of immunosuppressive therapy
* Participant has any of the following known untreated conditions; proliferative diabetic retinopathy, diabetic macular edema, macular degeneration or retinal vein occlusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 741 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meraf Eyassu, Study Director — Kyntra Bio
Locations (63):
- United States (61):
  - Research Center, Phoenix, Arizona
  - Research Center, Pine Bluff, Arkansas
  - Research Center, Chula Vista, California
  - Research Center, La Mesa, California
  - Research Center, Long Beach, California
  - Research Center, Los Angeles, California
  - Research Center, Northridge, California
  - Research Center, Ontario, California
  - Research Center, Roseville, California
  - Research Center, San Diego, California
  - Research Center, San Dimas, California
  - Research Center, San Gabriel, California
  - Research Center, Whittier, California
  - Research Center, Coral Springs, Florida
  - Research Center, Lauderdale Lakes, Florida
  - Research Center, Miami, Florida
  - Research Center, Pembroke Pines, Florida
  - Research Center, Tampa, Florida
  - Research Center, Albany, Georgia
  - Research Center, Meridian, Idaho
  - Research Center, Shreveport, Louisiana
  - Research Center, Springfield, Massachusetts
  - Research Center, Detroit, Michigan
  - Research Center, Pontiac, Michigan
  - Research Center, Brookhaven, Mississippi
  - Research Center, Columbus, Mississippi
  - Research Center, Gulfport, Mississippi
  - Research Center, Tupelo, Mississippi
  - Research Center, Creve Coeur, Missouri
  - Research Center, Kansas City, Missouri
  - Research Center, Saint Ann, Missouri
  - Research Center, St Louis, Missouri
  - Research Center, Portsmouth, New Hampshire
  - Research Center, North Brunswick, New Jersey
  - Research Center, Albuquerque, New Mexico
  - Research Center, Gallup, New Mexico
  - Research Center, College Point, New York
  - Research Center, New York, New York
  - Research Center, Charlotte, North Carolina
  - Research Center, Durham, North Carolina
  - Research Center, Greenville, North Carolina
  - Research Center, New Bern, North Carolina
  - Research Center, Raleigh, North Carolina
  - Research Center, Rocky Mount, North Carolina
  - Research Center, Columbus, Ohio
  - Research Center, Aiken, South Carolina
  - Research Center, Columbia, South Carolina
  - Research Center, Orangeburg, South Carolina
  - Research Center, Sumter, South Carolina
  - Research Center, Knoxville, Tennessee
  - Research Center, Nashville, Tennessee
  - Research Center, Arlington, Texas
  - Research Center, Edinburg, Texas
  - Research Center, Fort Worth, Texas
  - Research Center, Grand Prairie, Texas
  - Research Center, Houston, Texas
  - Research Center, Lubbock, Texas
  - Research Center, Mansfield, Texas
  - Research Center, San Antonio, Texas
  - Research Center, Alexandria, Virginia
  - Research Center, Shorewood, Wisconsin
- Puerto Rico (2):
  - Research Center, Caguas
  - Research Center, San Juan

REFERENCES:
- [Derived] Hamano T, Yamaguchi Y, Goto K, Martin S, Jiletcovici A, Dellanna F, Akizawa T, Barratt J. Risk Factors for Thromboembolic Events in Patients With Dialysis-Dependent CKD: Pooled Analysis of Four Global Roxadustat Phase 3 Trials. Adv Ther. 2024 Apr;41(4):1553-1575. doi: 10.1007/s12325-023-02728-2. Epub 2024 Feb 16. PMID 38363466
- [Derived] Barratt J, Dellanna F, Portoles J, Choukroun G, De Nicola L, Young J, Dimkovic N, Reusch M. Safety of Roxadustat Versus Erythropoiesis-Stimulating Agents in Patients with Anemia of Non-dialysis-Dependent or Incident-to-Dialysis Chronic Kidney Disease: Pooled Analysis of Four Phase 3 Studies. Adv Ther. 2023 Apr;40(4):1546-1559. doi: 10.1007/s12325-023-02433-0. Epub 2023 Feb 7. PMID 36749544
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive either roxadustat or epoetin alfa.
Groups:
- Roxadustat: Participants received roxadustat tablets, administered orally 3 times weekly (TIW). Initial roxadustat dose was based on the participant's average prescribed erythropoietin stimulating agent (ESA) dose in the 4 weeks (if on epoetin or darbepoetin or 8 weeks (if on Mircera®) prior to randomization. Dose adjustments were permitted to maintain a hemoglobin (Hb) level of approximately 11 grams (g)/deciliter (dL). The maximum roxadustat dose was 3.0 milligrams (mg)/kilogram (kg) per dose or 400 mg per administration (whichever was lower). The maximum treatment duration was 183.7 weeks.
- Epoetin Alfa: Participants on hemodialysis (HD) received epoetin alfa, administered intravenously (IV) TIW and participants on home HD or peritoneal dialysis (PD) received epoetin alfa, administered subcutaneously (SC). Initial epoetin alfa dose was based on the participant's average weekly prescribed ESA dose in 4 weeks prior to randomization if on epoetin or darbepoetin, and average monthly (4-week) prescribed ESA dose in 8 weeks prior to randomization if on Mircera®. In case of a change in route of administration from SC to IV (TIW), the initial dose of IV epoetin alfa was determined by the investigator per local standard of care (SOC). Dose adjustments followed the recommendations as per the approved country-specific product label (United States Package Insert [USPI] or Summary of Product Characteristics [SmPC]) or local SOC. The maximum treatment duration was 180.4 weeks.
Period: Overall Study
Arm/Group | Roxadustat | Epoetin Alfa
Started | 370 | 371
Received at Least 1 Dose of Study Drug | 370 | 370
Completed | 127 | 183
Not Completed | 243 | 188
Not completed — Death | 70 | 62
Not completed — Withdrawal by Subject | 41 | 29
Not completed — Kidney transplant | 31 | 39
Not completed — Physician Decision | 30 | 15
Not completed — Adverse Event | 27 | 9
Not completed — Lost to Follow-up | 6 | 3
Not completed — Lack of Efficacy | 6 | 1
Not completed — Protocol Violation | 4 | 0
Not completed — Other than specified | 28 | 30

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population included all randomized participants.
Groups:
- Roxadustat: Participants received roxadustat tablets, administered orally TIW. Initial roxadustat dose was based on the participant's average prescribed ESA dose in the 4 weeks (if on epoetin or darbepoetin or 8 weeks (if on Mircera®) prior to randomization. Dose adjustments were permitted to maintain a Hb level of approximately 11 g/dL. The maximum roxadustat dose was 3.0 mg/kg per dose or 400 mg per administration (whichever was lower). The maximum treatment duration was 183.7 weeks.
- Epoetin Alfa: Participants on HD received epoetin alfa, administered IV TIW and participants on home HD or PD received epoetin alfa, administered SC. Initial epoetin alfa dose was based on the participant's average weekly prescribed ESA dose in 4 weeks prior to randomization if on epoetin or darbepoetin, and average monthly (4-week) prescribed ESA dose in 8 weeks prior to randomization if on Mircera®. In case of a change in route of administration from SC to IV (TIW), the initial dose of IV epoetin alfa was determined by the investigator per local SOC. Dose adjustments followed the recommendations as per the approved country-specific product label (USPI or SmPC) or local SOC. The maximum treatment duration was 180.4 weeks.
- Total: Total of all reporting groups
Arm/Group | Roxadustat | Epoetin Alfa | Total
Number analyzed (Participants) | 370 | 371 | 741
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 253 | 246 | 499
  >=65 years | 117 | 125 | 242
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 156 | 339
  Male | 187 | 215 | 402
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 137 | 129 | 266
  Not Hispanic or Latino | 233 | 242 | 475
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 165 | 184 | 349
  Race: Black/African American | 158 | 156 | 314
  Race: Asian | 21 | 15 | 36
  Race: American Indian/Alaskan Native | 10 | 7 | 17
  Race: Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Race: Other | 15 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: US (FDA) Submission: Mean Hb Change From Baseline to The Average Level During The Evaluation Period (Weeks 28 to 52), Regardless of Rescue Therapy
Description: Hb values under the influence of rescue therapy were not censored in the analysis. Rescue therapy for roxadustat treated participants was defined as recombinant erythropoietin or analogue (ESA) or red blood cell (RBC) transfusion, and rescue therapy for epoetin alfa treated participants was defined as RBC transfusion. Baseline Hb was defined the mean of up to 4 last central lab values prior to the first dose of study treatment. The intermittent missing Hb data was imputed for each treatment relying on non-missing data from all participants within each treatment group using the Monte Carlo Markov Chain (MCMC) imputation model, Monotone missing data were imputed by regression from its own treatment group.
Time Frame: Baseline (Day 1, Week 0), Weeks 28 to 52
Population: ITT Population included all randomized participants.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 370 | 371
g/dL
  Baseline | 10.30 (0.661) | 10.31 (0.656)
  Change at Weeks 28 to 52 | 0.39 (0.934) | -0.09 (0.838)
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Treatment comparison was made using the multiple imputation (MI) strategy by combining the results of analysis of covariance (ANCOVA) model with baseline Hb as a covariate, and treatment, ESA dependent incident dialysis within ≤4 months vs. >4 months of starting dialysis when randomized, and other randomization stratification factors except mean qualifying screening hemoglobin (≤10.5 vs. >10.5 g/dL) as fixed effects; Test type: Non-Inferiority — Non-inferiority was established if the 2-sided 95% confidence interval (CI) for the treatment difference in least square (LS) means from MI ANCOVA model between the 2 treatment groups lay entirely above -0.75 g/dL; p < 0.0001, ANCOVA; ANCOVA with MI; LS Mean Difference = 0.48, 95% CI 2-sided [0.365 to 0.591], Standard Error of Mean 0.058

2. Primary Outcome: Ex-U.S. Submission: Mean Hb Change From Baseline to the Average Weeks 28 to 36, Without Having Received Rescue Therapy Within 6 Weeks Prior to and During This 8-Week Evaluation Period for Participants Enrolled Under the Original Protocol
Description: Hb values under the influence of rescue therapy were censored up to 6 weeks in the analysis. Rescue therapy for roxadustat treated participants was defined as recombinant erythropoietin or analogue (ESA) or RBC transfusion, and rescue therapy for epoetin alfa treated participants was defined as RBC transfusion. Baseline Hb was defined the mean of up to 4 last central lab values prior to the first dose of study treatment.
Time Frame: Baseline (Day 1, Week 0), Weeks 28 to 36
Population: Per protocol set (PPS) population included all participants in full analysis set (FAS) population (all randomized participants who received at least 1 dose of study drug and had at least 1 postdose Hb assessment) who received at least 8 weeks of treatment and were without major protocol violations. 'Overall number of participants analyzed'=participants evaluable for this outcome measure. 'Number analyzed'=participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 303 | 324
g/dL
  Baseline | 10.33 (0.639) | 10.35 (0.614)
  Change at Weeks 28 to 36: number analyzed (Participants) | 263 | 293
  Change at Weeks 28 to 36 | 0.54 (1.022) | -0.03 (0.897)
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Treatment comparison was made using a mixed model of repeated measures (MMRM) with baseline Hb as a covariate, and treatment, visit, visit-by-treatment interaction, ESA dependent incident dialysis within ≤4 months vs. >4 months of starting dialysis when randomized, and randomization stratification factors except mean qualifying screening Hb (≤10.5 vs. >10.5 g/dL) as fixed effects; Test type: Non-Inferiority — The non-inferiority was established when the 2-sided 95% CI for the difference of LS means between the 2 treatment groups using the MMRM model lay entirely above -0.75 g/dL; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 0.55, 95% CI 2-sided [0.404 to 0.687], Standard Error of Mean 0.072

3. Secondary Outcome: US (FDA Submission): Hb Responder Rate- Percentage of Participants With Mean Hb Level ≥10.0 g/dL Averaged Over Weeks 28 to 52, Regardless of Rescue Therapy
Description: Hb values under the influence of rescue therapy were not censored in the analysis. Rescue therapy for roxadustat treated participants was defined as recombinant erythropoietin or analogue (ESA) or RBC transfusion, and rescue therapy for epoetin alfa treated participants was defined as RBC transfusion.
Time Frame: Weeks 28 to 52
Population: FAS population included all randomized participants who received at least 1 dose of study drug and had at least 1 postdose Hb assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 369 | 370
percentage of participants | 66.1 | 58.6
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; For the difference of responder rates between 2 treatment groups, the CI analyzed was from the Miettinen & Nurminen approach adjusting for randomization stratification factors; Test type: Non-Inferiority — Non-inferiority was established if the lower bound of the 2-sided 95% CI for the treatment difference for the responder rates (roxadustat minus epoetin alfa) calculated based on the Miettinen & Nurminen approach, adjusting for stratification factors, was greater than -15%; Responder Rate Difference = 7.6, 95% CI 2-sided [0.9 to 14.3]

4. Secondary Outcome: Ex-U.S. Submission: Hb Responder Rate- Percentage of Participants With Mean Hb 10.0 to 12.0 g/dL Averaged Over Weeks 28 to 36, Censoring for Rescue Therapy
Description: Hb values under the influence of a rescue therapy were censored up to 6 weeks in the analysis. Rescue therapy for roxadustat treated participants was defined as recombinant erythropoietin or analogue (ESA) or RBC transfusion, and rescue therapy for epoetin alfa treated participants was defined as RBC transfusion.
Time Frame: Weeks 28 to 36
Population: The PPS population included all participants in the FAS population (all randomized participants who received at least 1 dose of study drug and had at least 1 postdose Hb assessment) who received at least 8 weeks of treatment, had at least 1 valid postdose Hb assessment and were without major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 334 | 352
percentage of participants | 64.1 | 60.8
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Responder Rate Difference = 2.7, 95% CI 2-sided [-4.3 to 9.7]

5. Secondary Outcome: Change From Baseline in Low-Density Lipoprotein (LDL) Cholesterol Averaged Over Weeks 12 to 28
Description: Baseline LDL Cholesterol was defined as the last available value prior to the first dose of study treatment.
Time Frame: Baseline (Day 1, Week 0), Weeks 12 to 28
Population: FAS population included all randomized participants who received at least 1 dose of study drug and had at least 1 postdose Hb assessment. Here, 'Number analyzed' signifies participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 369 | 370
mg/dL
  Baseline | 84.53 (34.009) | 84.45 (34.124)
  Change at Weeks 12 to 28: number analyzed (Participants) | 327 | 354
  Change at Weeks 12 to 28 | -13.70 (23.068) | 1.23 (22.389)
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Treatment comparison was made using a MMRM with baseline as a covariate, and treatment, visit, visit-by-treatment interaction, ESA dependent incident dialysis within ≤4 months vs. >4 months of starting dialysis when randomized, and randomization stratification factors as fixed effects; Test type: Superiority — Superiority was declared if the upper bound of the 2-sided 95% CI of the difference between roxadustat and epoetin alfa (roxadustat - epoetin alpha) was less than 0; p < 0.0001, Mixed Models Analysis; Least Square Mean Difference = -14.67, 95% CI 2-sided [-17.640 to -11.695], Standard Error of Mean 1.514

6. Secondary Outcome: Change From Baseline in Hb Levels Averaged Over Weeks 18 to 24 Regardless of Rescue Therapy in Participants Whose Baseline High Sensitivity C-Reactive Protein (Hs-CRP)> Upper Limit of Normal (ULN)
Description: Hb values under the influence of rescue therapy were not censored in the analysis. Rescue therapy for roxadustat treated participants was defined as recombinant erythropoietin or analogue (ESA) or RBC transfusion, and rescue therapy for epoetin alfa treated participants was defined as RBC transfusion. Baseline Hb was defined the mean of up to 4 last central lab values prior to the first dose of study treatment. The intermittent missing Hb data was imputed for each treatment relying on non-missing data from all participants within each treatment group using the MCMC imputation model, Monotone missing data were imputed by regression from its own treatment group.
Time Frame: Baseline (Day 1, Week 0), Weeks 18 to 24
Population: FAS population included all randomized participants who received at least 1 dose of study drug and had at least 1 postdose Hb assessment. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 189 | 176
g/dL
  Baseline | 10.30 (0.616) | 10.24 (0.630)
  Change at Weeks 18-24 | 0.61 (1.020) | -0.03 (0.940)
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Treatment comparison was made using the MI strategy by combining the results of ANCOVA model with baseline Hb as a covariate, and treatment, ESA dependent incident dialysis within ≤4 months vs. >4 months of starting dialysis when randomized, and other randomization stratification factors except mean qualifying screening Hb (≤10.5 vs. >10.5 g/dL) as fixed effects; Test type: Non-Inferiority — The non-inferiority margin was fixed as a difference of -0.75; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; ANCOVA with MI; LS Mean Difference = 0.69, 95% CI 2-sided [0.503 to 0.869], Standard Error of Mean 0.093

7. Secondary Outcome: Average Monthly IV Iron Use Per Patient-Exposure-Month (PEM) During Weeks 28 to 52
Description: Monthly iron use for each participant= Total IV iron in mg / [(last dose date - first dose date of study medication in the period)+1]/ 28.
Time Frame: Weeks 28 to 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/PEM
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 286 | 319
mg/PEM | 17.07 (53.375) | 37.02 (106.778)
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Treatment comparison was made using an ANCOVA model with baseline iron repletion status, treatment, ESA dependent incident dialysis within ≤4 months vs. >4 months of starting dialysis when randomized, and randomization stratification factors as fixed effects; Test type: Superiority; p = 0.00091, Rank ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -20.14, 95% CI 2-sided [-33.842 to -6.445], Standard Error of Mean 6.975

8. Secondary Outcome: Time to First RBC Transfusion
Description: Median time to event (weeks) was calculated using Kaplan Meier Survival Estimates.
Time Frame: Baseline (Day 1, Week 0) up to last dose of study drug (maximum treatment duration was 183.7 weeks for roxadustat and 180.4 weeks for epoetin alfa)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 369 | 370
weeks | NA [NA to NA] — Due to smaller number of participants with an event (any use of RBC transfusion), median and 95% CI could not be calculated. | NA [NA to NA] — Due to smaller number of participants with an event (any use of RBC transfusion), median and 95% CI could not be calculated.
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Analysis was done using a Cox Proportional Hazards model adjusting for baseline Hb and other stratification factors except mean qualifying screening Hb (≤10.5 vs. >10.5 g/dL) as fixed effects; Test type: Non-Inferiority — The non-inferiority margin for the difference between groups was 1.8; p = 0.0337, Cox Proportional Hazards model; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.466 to 0.970]

9. Secondary Outcome: Change From Baseline in Mean Arterial Pressure (MAP) Averaged Over Weeks 20 to 28
Description: Baseline MAP was defined as the mean of values obtained within 6 weeks prior to the first dose of study treatment.
Time Frame: Baseline (Day 1, Week 0), Weeks 20 to 28
Population: FAS population included all randomized participants who received at least 1 dose of study drug and had at least 1 postdose Hb assessment. Here, 'Number analyzed' signifies participants evaluable for this outcome measure at specified timepoints.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 369 | 370
millimeters of mercury (mmHg)
  Baseline | 101.41 (12.591) | 100.34 (12.350)
  Change at Weeks 20 to 28: number analyzed (Participants) | 304 | 338
  Change at Weeks 20 to 28 | 0.46 (10.933) | 0.04 (10.489)
Statistical Analysis 1: Comparison: Roxadustat vs Epoetin Alfa; Treatment comparison was made using MMRM with baseline as a covariate, and treatment, visit, visit-by-treatment interaction, ESA dependent incident dialysis within ≤4 months vs. >4 months of starting dialysis when randomized, and randomization stratification factors as fixed effects; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.3500, Mixed Models Analysis; LS Mean Difference = 0.69, 95% CI 2-sided [-0.760 to 2.142], Standard Error of Mean 0.739

10. Secondary Outcome: Time to First Exacerbation of Hypertension During Weeks 28 to 52
Description: An exacerbation of hypertension was defined as increase from baseline of ≥20 mmHg in systolic blood pressure (sBP) and sBP ≥170 mmHg or an increase from baseline of ≥15 mmHg in diastolic blood pressure (dBP) and dBP ≥100 mmHg. Median time to event (weeks) was calculated using Kaplan Meier Survival Estimates.
Time Frame: Weeks 28 to 52
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 369 | 370
weeks | NA [NA to NA] — Due to smaller number of participants with an event (exacerbation hypertension), median and 95% CI could not be calculated. | NA [NA to NA] — Due to smaller number of participants with an event (exacerbation hypertension), median and 95% CI could not be calculated.

11. Secondary Outcome: Change From Baseline in Short Form 36 (SF-36) Version 2 Physical Functioning Subscore and Vitality Subscore at Weeks 12 to 28
Description: The SF-36 V2 consists of 36 questions covering 8 health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical problems (4 items), role limitations due to emotional problems (3 items), general health perceptions (5 items), mental health (5 items), social function (2 items), and vitality (4 items). The physical functioning subscore and vitality subscore are reported. Each scale was transformed into 0-100 score, with higher scores indicating better health status. Baseline score was defined as the last physical functioning value or vitality value, as applicable, prior to the first dose of study drug.
Time Frame: Baseline (Day 1, Week 0), Weeks 12 to 28
Population: FAS Population included all randomized/enrolled participants who received at least 1 dose of study drug and had baseline and at least 1 postdose Hb assessment. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for this outcome measure at specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roxadustat | Epoetin Alfa
Number analyzed (Participants) | 368 | 369
score on a scale
  Physical functioning subscore: Baseline | 38.55 (11.202) | 39.63 (11.368)
  Physical functioning subscore: Change at Weeks 12 to 28: number analyzed (Participants) | 326 | 352
  Physical functioning subscore: Change at Weeks 12 to 28 | -0.15 (7.443) | -0.20 (6.380)
  Vitality subscore: Baseline | 51.65 (10.111) | 51.27 (9.841)
  Vitality subscore: Change at Weeks 12 to 28: number analyzed (Participants) | 326 | 352
  Vitality subscore: Change at Weeks 12 to 28 | -0.92 (7.007) | 0.30 (7.041)

ADVERSE EVENTS:
Time Frame: Baseline (Day 1, Week 0) up to 28 days after the last dose of study drug (maximum treatment duration was 183.7 weeks for roxadustat and 180.4 weeks for epoetin alfa). Mortality presented is for the timeframe of Baseline (Day 1, Week 0) up to end of treatment (maximum treatment duration was 183.7 weeks for roxadustat and 180.4 weeks for epoetin alfa).
Description: The Safety population included all randomized participants who received at least 1 dose of study medication.
Arm/Group | Roxadustat | Epoetin Alfa
All-Cause Mortality (participants affected / at risk) | 70/370 | 62/370
Serious Adverse Events (participants affected / at risk) | 242/370 | 248/370
Other Adverse Events (participants affected / at risk) | 286/370 | 292/370
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roxadustat (N=370) | Epoetin Alfa (N=370)
Anaemia (Blood and lymphatic system disorders) | 16 | 20
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 6
Acute myocardial infarction (Cardiac disorders) | 31 | 26
Cardiac failure congestive (Cardiac disorders) | 23 | 23
Cardiac arrest (Cardiac disorders) | 20 | 23
Coronary artery disease (Cardiac disorders) | 11 | 12
Atrial fibrillation (Cardiac disorders) | 9 | 11
Cardiorespiratory arrest (Cardiac disorders) | 8 | 9
Angina unstable (Cardiac disorders) | 7 | 3
Myocardial infarction (Cardiac disorders) | 5 | 3
Angina pectoris (Cardiac disorders) | 4 | 6
Bradycardia (Cardiac disorders) | 4 | 4
Pulseless electrical activity (Cardiac disorders) | 4 | 1
Cardiogenic shock (Cardiac disorders) | 4 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 10 | 16
Colitis (Gastrointestinal disorders) | 4 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 4
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 4
Gastric ulcer (Gastrointestinal disorders) | 0 | 4
Non-cardiac chest pain (General disorders) | 17 | 10
Asthenia (General disorders) | 3 | 7
Death (General disorders) | 1 | 4
Pneumonia (Infections and infestations) | 30 | 39
Sepsis (Infections and infestations) | 18 | 23
Septic shock (Infections and infestations) | 10 | 7
Cellulitis (Infections and infestations) | 9 | 15
Urinary tract infection (Infections and infestations) | 8 | 6
Gastroenteritis (Infections and infestations) | 8 | 3
Arteriovenous fistula site infection (Infections and infestations) | 7 | 1
Influenza (Infections and infestations) | 6 | 6
Staphylococcal bacteraemia (Infections and infestations) | 6 | 6
Osteomyelitis (Infections and infestations) | 3 | 12
Gangrene (Infections and infestations) | 4 | 8
Diverticulitis (Infections and infestations) | 4 | 6
Bronchitis (Infections and infestations) | 4 | 4
Bacteraemia (Infections and infestations) | 3 | 6
Arteriovenous graft site infection (Infections and infestations) | 3 | 4
Clostridium difficile colitis (Infections and infestations) | 3 | 4
Device related infection (Infections and infestations) | 2 | 5
Staphylococcal sepsis (Infections and infestations) | 2 | 4
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 11 | 11
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 10 | 7
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 8 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 7
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 3 | 4
Femur fracture (Injury, poisoning and procedural complications) | 2 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 25 | 25
Fluid overload (Metabolism and nutrition disorders) | 24 | 27
Hypoglycaemia (Metabolism and nutrition disorders) | 7 | 9
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 | 4
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Syncope (Nervous system disorders) | 7 | 12
Seizure (Nervous system disorders) | 7 | 8
Encephalopathy (Nervous system disorders) | 6 | 5
Cerebrovascular accident (Nervous system disorders) | 4 | 5
Metabolic encephalopathy (Nervous system disorders) | 5 | 11
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 5
Mental status changes (Psychiatric disorders) | 5 | 8
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 15 | 26
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 12
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 15
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Diabetic foot (Skin and subcutaneous tissue disorders) | 3 | 4
Hypotension (Vascular disorders) | 18 | 19
Deep vein thrombosis (Vascular disorders) | 9 | 5
Hypertension (Vascular disorders) | 6 | 4
Peripheral ischaemia (Vascular disorders) | 5 | 0
Hypertensive crisis (Vascular disorders) | 4 | 3
Aortic stenosis (Vascular disorders) | 0 | 4
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 2
Acute left ventricular failure (Cardiac disorders) | 1 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 3
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 2
Cardiovascular disorder (Cardiac disorders) | 1 | 1
Chronic left ventricular failure (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Mitral valve stenosis (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 2 | 2
Palpitations (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 1
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 3
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 2 | 2
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 2
Hyperparathyroidism tertiary (Endocrine disorders) | 2 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 3
Colitis ischaemic (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Diabetic gastroparesis (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Diverticulum (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1
Erosive duodenitis (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 2 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 2
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0
Oesophageal polyp (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 3 | 0
Pancreatitis acute (Gastrointestinal disorders) | 3 | 3
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Reactive gastropathy (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 3
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Tongue dysplasia (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 1
Uraemic gastropathy (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Chest pain (General disorders) | 3 | 2
Complication associated with device (General disorders) | 3 | 1
Drowning (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 1
Hypothermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 3 | 0
Oedema peripheral (General disorders) | 2 | 1
Pain (General disorders) | 0 | 1
Pelvic mass (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 2 | 0
Pyrexia (General disorders) | 3 | 1
Sudden cardiac death (General disorders) | 2 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 3 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 2
Jaundice (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1
Kidney transplant rejection (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 2 | 0
Abscess limb (Infections and infestations) | 1 | 1
Abscess oral (Infections and infestations) | 0 | 1
Abscess soft tissue (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 3 | 3
Appendicitis perforated (Infections and infestations) | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 1
Cardiac valve vegetation (Infections and infestations) | 0 | 1
Cellulitis staphylococcal (Infections and infestations) | 0 | 1
Citrobacter sepsis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 2 | 1
Endocarditis (Infections and infestations) | 1 | 1
Endocarditis bacterial (Infections and infestations) | 1 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Extradural abscess (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 0 | 1
Gastroenteritis clostridial (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 1
Graft infection (Infections and infestations) | 2 | 0
Haemophilus infection (Infections and infestations) | 0 | 1
Implant site infection (Infections and infestations) | 0 | 1
Infected seroma (Infections and infestations) | 1 | 1
Infectious colitis (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 1 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 3 | 1
Ludwig angina (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0
Osteomyelitis acute (Infections and infestations) | 0 | 2
Osteomyelitis bacterial (Infections and infestations) | 0 | 1
Osteomyelitis bacterial (Infections and infestations) | 1 | 1
Pelvic abscess (Infections and infestations) | 1 | 1
Perirectal abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 2 | 3
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 3
Postoperative wound infection (Infections and infestations) | 0 | 2
Proteus infection (Infections and infestations) | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 | 0
Septic embolus (Infections and infestations) | 1 | 0
Septic phlebitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 3
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal infection (Infections and infestations) | 1 | 0
Subacute endocarditis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Urinary tract infection fungal (Infections and infestations) | 0 | 1
Vascular access site infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Vulval abscess (Infections and infestations) | 1 | 0
Vulval cellulitis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 1
Wound sepsis (Infections and infestations) | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 1
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 | 1
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous graft site haematoma (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 2 | 2
Arteriovenous graft site stenosis (Injury, poisoning and procedural complications) | 0 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 2
Gun shot wound (Infections and infestations) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 2
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 2 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular access malfunction (Injury, poisoning and procedural complications) | 2 | 0
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 2
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Troponin increased (Investigations) | 2 | 0
Calciphylaxis (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Brown tumour (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Uraemic myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Large granular lymphocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm of thorax (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Nasopharyngeal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Allodynia (Nervous system disorders) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 1
Ataxia (Nervous system disorders) | 1 | 0
Brain injury (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Cerebellar stroke (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Facial paralysis (Nervous system disorders) | 1 | 2
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 2 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 1
Ischaemic strok (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 3 | 3
Sciatica (Nervous system disorders) | 2 | 0
Thalamic infarction (Nervous system disorders) | 0 | 1
Thoracic outlet syndrome (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 3
Tremor (Nervous system disorders) | 0 | 1
Acute psychosis (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Anxiety disorder (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 2 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 3
Major depression (Psychiatric disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 3 | 2
End stage renal disease (Renal and urinary disorders) | 1 | 2
Haematuria (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Renal haemorrhage (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Renal mass (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Accelerated hypertension (Vascular disorders) | 2 | 2
Arteriosclerosis (Vascular disorders) | 2 | 0
Brachiocephalic vein occlusion (Vascular disorders) | 0 | 1
Dry gangrene (Vascular disorders) | 1 | 3
Essential hypertension (Vascular disorders) | 1 | 2
Extremity necrosis (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypertensive emergency (Vascular disorders) | 3 | 3
Hypovolaemic shock (Vascular disorders) | 0 | 2
Iliac vein occlusion (Vascular disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 1
Malignant hypertension (Vascular disorders) | 0 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 1
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 2 | 3
Secondary hypertension (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 2 | 2
Steal syndrome (Vascular disorders) | 2 | 0
Superior vena cava stenosis (Vascular disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Venous stenosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Roxadustat (N=370) | Epoetin Alfa (N=370)
Anaemia (Blood and lymphatic system disorders) | 28 | 41
Tachycardia (Cardiac disorders) | 20 | 19
Bradycardia (Cardiac disorders) | 11 | 19
Nausea (Gastrointestinal disorders) | 63 | 60
Vomiting (Gastrointestinal disorders) | 60 | 55
Diarrhoea (Gastrointestinal disorders) | 54 | 69
Constipation (Gastrointestinal disorders) | 44 | 48
Abdominal pain (Gastrointestinal disorders) | 32 | 30
Abdominal pain upper (Gastrointestinal disorders) | 19 | 16
Non-cardiac chest pain (General disorders) | 24 | 32
Pyrexia (General disorders) | 32 | 33
Asthenia (General disorders) | 25 | 15
Oedema peripheral (General disorders) | 22 | 34
Peripheral swelling (General disorders) | 16 | 26
Face oedema (General disorders) | 10 | 19
Upper respiratory tract infection (Infections and infestations) | 43 | 40
Pneumonia (Infections and infestations) | 19 | 22
Urinary tract infection (Infections and infestations) | 24 | 26
Viral upper respiratory tract infection (Infections and infestations) | 26 | 26
Bronchitis (Infections and infestations) | 22 | 25
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 53 | 71
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 29 | 32
Fall (Injury, poisoning and procedural complications) | 36 | 53
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 24 | 27
Contusion (Injury, poisoning and procedural complications) | 14 | 20
Vascular graft complication (Injury, poisoning and procedural complications) | 9 | 22
Hyperkalaemia (Metabolism and nutrition disorders) | 38 | 43
Fluid overload (Metabolism and nutrition disorders) | 17 | 25
Hypoglycaemia (Metabolism and nutrition disorders) | 20 | 21
Iron deficiency (Metabolism and nutrition disorders) | 12 | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 49 | 58
Back pain (Musculoskeletal and connective tissue disorders) | 37 | 39
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 37
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 | 25
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15 | 20
Headache (Nervous system disorders) | 42 | 40
Dizziness (Nervous system disorders) | 24 | 30
Anxiety (Psychiatric disorders) | 16 | 20
Insomnia (Psychiatric disorders) | 15 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 49 | 69
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 56 | 64
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 21
Hypertension (Vascular disorders) | 59 | 44
Hypotension (Vascular disorders) | 27 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The multisite consortium can publish any time after the data is collected and analyzed by FibroGen.

The investigator can only publish after the multisite consortium publishes (or tries to publish and fails).

FibroGen has 60 days to review a publication and can extend the embargo up to an additional 120 days (or 180 total).

DOCUMENTS (2):
  • Study Protocol (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT02273726/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT02273726/SAP_001.pdf